CLINICAL TRIAL: NCT03239652
Title: Safety and Efficacy of Prostatic Artery Embolization Therapy in Symptomatic Benign Prostatic Hyperplasia
Brief Title: Taiwan ACE Beads for Embolization Therapy in Symptomatic Benign Prostatic Hyperplasia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cheng-Kung University Hospital (Other)
Collaborators: The Industrial Technology Research Institute (Other); National Cheng Kung University (Other); National Research Program for Biopharmaceuticals, Taiwan (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A-BR-105-055
Record Dates: First submitted 2017-07-25; First posted 2017-08-04 (Actual); Last update posted 2019-10-17 (Actual); Status verified 2019-08

CONDITIONS: Lower Urinary Tract Symptom; Benign Prostatic Hyperplasia (BPH)
Keywords: Microsphere; Transcatheter Arterial chemo-embolization
MeSH Terms: conditions — Lower Urinary Tract Symptoms; Prostatic Hyperplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Taiwan ACE Beads microspheres (Experimental): The maximum use of dosage will not exceed 100 milligrams. The embolization procedure usually lasts less than an hour.
  Interventions: Device: Taiwan ACE Beads

INTERVENTIONS:
Device: Taiwan ACE Beads — Similar with conventional Transcatheter Arterial chemo-embolization, radiologist use Taiwan ACE Beads instead of Gelfoam or polyvinyl alcohol.

SUMMARY:
In this proposal, the investigators plan to conduct a clinical trial to validate the efficacy and safety of microspheres (T-ACE Beads).

DETAILED DESCRIPTION:
T-ACE Beads can be used for prostatic arterial embolization safely and efficiently. Furthermore, investigator's microspheres has advantageous characteristics in biodegradability, drug delivery capability, and cost-effectiveness. After the clinical trial, we anticipate introducing a new microsphere for Lower Urinary Tract Symptom/Benign prostatic hyperplasia patients, which is beneficial to the participants in precise medicine as well as in the pharmaceutical and medical device industry.

ELIGIBILITY:
Inclusion Criteria:

A. Men ≥ 50 years of age. Healthy patients or volunteers without diagnosis of Lower urinary tract symptoms (LUTS) / Benign prostatic hyperplasia (BPH) will not be included.

B. Patients diagnosed of LUTS / BPH，International Prostate Symptom Score > 12 with mild to severe symptom of LUTS.

C. Prostate volume > 50 mL.

D. Urinary flow rate <15 mL / sec.

E. Ineffectiveness after 6 months of previous medical treatment, or the side effects are too difficult to tolerate.

Exclusion Criteria:

If patients meet any of the following criteria they may not be entered into the study:

A. Major pelvic disease, or other malignancies.

B. Prostate specific antigen of serum > 10 ng/mL, malignant tumor not yet rule out (prostate specific antigen PSA>10 ng/mL).

C. Had Prostate surgery.

D. Chronic bacterial prostatitis.

E. Renal dysfunction or bladder diverticulum stones caused by prostate disease obstruction.

F. Main organs (heart, lung, liver, kidney) dysfunction who are not eligible for clinical trials under physicians' consideration.

G. White Blood Cell< 2000 or Severe thrombocytopenia（Platelet count <50,000/μL)，or blood coagulation abnormalities uncorrectable .

H. Unable to follow-up by MRI 3 times.

I. Unable to follow-up by ultrasound or CT scan.

J. Unwilling to sign a written informed consent form.

K. Allergic to Iodine or other injections.

L. Acute bacterial prostatitis.

M. Patients with active urinary tract infections or recurrent urinary tract infections (>2/years), prostatitis, or interstitial cystitis.

N. Cases of biopsy proven prostate, bladder, or urethral cancer.

O. Patients with glomerular filtration rates less than 40 who are not already on dialysis.

P. Patients with bilateral internal iliac arterial occlusion.

Q. Patients with causes of bladder obstruction not due to BPH (eg urethral stricture, bladder neck contraction, etc).

R. Patients with neurogenic or bladder atonia.

S. Patients where embolization is not possible distal to collateral vessels feeding non-prostatic tissue.

T. Patients with major neurologic illnesses which could have symptoms that may be similar to or confused for BPH (eg multiple sclerosis, Shy-Drager syndrome, spinal cord injury, etc.).

U. Patients with urethral stents.

V. Other than hemorrhoidectomy or pelvic irradiation, patients who have undergone prior rectal surgery.

W. Patients who have started or changed their dosage of alpha blockers or 5-alpha reductase inhibitors in the month prior to prostatic artery embolization.

X. Allergic to pharmaceutical excipients related to Microspheres.

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Patients Survival (Safety) | An average of 12 weeks.
  Survival rate was evaluated since treatment day until the date of death or final observation.

SECONDARY OUTCOMES:
Change on Patient's Symptoms | Before treatment, one and three months after treatment
  Change on patients' International Prostate Symptom Score (IPSS)
Change on Prostate Volume | Before treatment, one and three months after treatment.
  Prostate volume measured using MRI
Change in serum Prostate Specific Antigen (PSA) concentration | Before treatment, one and three months after treatment.
  Measurement of Prostate Specific Antigen in patients undergoing this treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Yuh-Shyan Tsai, MD, Principal Investigator — Department of Urology, National Cheng Kung University Hospital, College of medicine, National Cheng Kung University, Tainan 70403, Taiwan
Locations (1):
- National Cheng Kung University Hospital, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Liu YS, Lin XZ, Tsai HM, Tsai HW, Chen GC, Chen SF, Kang JW, Chou CM, Chen CY. Development of biodegradable radiopaque microsphere for arterial embolization-a pig study. World J Radiol. 2015 Aug 28;7(8):212-9. doi: 10.4329/wjr.v7.i8.212. PMID 26339465
- [Result] Noor A, Fischman AM. Prostate Artery Embolization as a New Treatment for Benign Prostate Hyperplasia: Contemporary Status in 2016. Curr Urol Rep. 2016 Jul;17(7):51. doi: 10.1007/s11934-016-0608-0. PMID 27146488